CLINICAL TRIAL: NCT03206684
Title: A Prospective, Open, Randomized, Controlled Clinical Study to Evaluate the Efficacy and Safety of PEG-rhG-CSF in Reducing Neutropenia in Patients With Cervical Cancer
Brief Title: To Evaluate the Efficacy and Safety of PEG-rhG-CSF（Jinyouli®） in Reducing Neutropenia in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-CC-01
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF (Experimental): PEG-rhG-CSF single-dose was administered subcutaneously 48h after chemotherapy，with patients' weight ≥ 45kg were given 6mg once per chemotherapy cycle, weight <45kg were given 3mg once per chemotherapy cycle.
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF (Active Comparator): rhG-CSF was daily administered subcutaneously 48h after chemotherapy，weight≥45kg were given 300μg/d, weight<45kg were given 150μg/d,continuous injection for 3-5 days until the absolute neutrophils count≥2×10^9/L.
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF single-dose was administered subcutaneously 48h after chemotherapy，weight ≥ 45kg were given 6mg once per chemotherapy cycle, weight <45kg were given 3mg once per chemotherapy cycle.
  Other Names: PEG-rhG-CSF single-dose administered
  Arms: PEG-rhG-CSF
Drug: rhG-CSF — rhG-CSF was administered subcutaneously 48h after chemotherapy，weight≥45kg were given 300μg/d, weight<45kg were given 150μg/d,continuous injection for 3-5 days until the absolute neutrophils count≥2×10^9/L.
  Other Names: rhG-CSF daily administered
  Arms: rhG-CSF

SUMMARY:
A Prospective, open, randomized, controlled clinical study to evaluate the efficacy and safety of PEG-rhG-CSF(PEGylated recombinant human granulocyte stimulating factor injection) in reducing neutropenia during TP(docetaxel+cisplatin) regiment simultaneous radiochemotherapy and adjuvant chemotherapy in patients with cervical cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤70 years old;
2. Cervical cancer patients diagnosed by histopathology;
3. Need to receive multi-cycle radical concurrent radiochemotherapy;
4. FN risk > 20% if rhG-CSF was not accepted; High risk factors associated with FN and planed to use the same protocol in subsequent cycles(docetaxel+cisplatin regimen)；
5. Performance status score(KPS)≥70;
6. No obvious blood system disease,absolute neutrophil count（ANC）≥ 1.5×10^9/L, platelet count≥80×10^9 /L, hemoglobin（Hb）≥75 g/L, and no bleeding tendency;
7. The patient signs the informed consent.

Exclusion Criteria:

1. With infection difficult to control, or received system antibiotic treatment within 72 h before chemotherapy;
2. Any bone marrow abnormalities and other hematopoietic ;
3. Had received bone marrow or hematopoietic stem cell transplantation within 3 months;
4. with other malignancies not cure, or with brain metastases;
5. Liver function tests:total bilirubin(TBIL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were all ≥2.5 times normal upper limit.
6. Renal function tests: serum creatinine (Cr)> 1.5 times normal upper limit;
7. Allergic to the drugs or other genetic engineering biological products from Escherichia coli;
8. Suffering from mental or neurological disorders;
9. Investigator think it is not suitable for recruiting.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of III/IV neutropenia | 3 months
  The incidence of III/IV neutropenia in each chemotherapy cycle

SECONDARY OUTCOMES:
Incidence of FN | 3 months
  Incidence of febrile neutropenia (FN) in each chemotherapy cycle
Proportion of chemotherapy dose adjustment | 3 months
  Proportion of chemotherapy dose adjustment due to neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Mei Shi, MD, Principal Investigator — Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China